CLINICAL TRIAL: NCT05343104
Title: Osteoarthrosis on 7.0T Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Director and Clinical Professor, Chinese PLA General Hospital
Other Study IDs: Osteoarthrosis-ChinaPLAGH
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: MRI; Osteoarthrosis
Keywords: MRI; Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Patients recruited will receive Magnetic resonance imaging.

SUMMARY:
This clinical trial studies the use of 7-Tesla (7T)and 3T magnetic resonance imaging (MRI) in detecting osteoarthrosis. 7T MRI has increased detection sensitivity, including more accurate lesion delineation, higher inter-rater agreement. Diagnostic procedures such as 7T MRI may help ultimately improved diagnostic and therapies confidence to inform decision making than standard 3T MRI.

DETAILED DESCRIPTION:
7T MRI increased detection sensitivity, attain superior anatomic resolution, higher spatial and spectral specificity of advanced quantitative techniques, and shorter scan times than 3T MRI. When applied clinically, these benefits translate to increased detection sensitivity, and ultimately improved diagnostic and therapies confidence to inform decision making. This study aim to detect the image characteristics and diagnostic accuracy of osteoarthrosis on 7T MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 and ≤80
* Having no contraindications against MRI
* Clinically stable

Exclusion Criteria:

* Age#18 or #80
* Pregnancy and other contraindication to MRI scan
* Informed consent not obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with clinical diagnosis of patellar chondromalacia were continuously included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The thickness of the cartilage of patellar on 7T MRI scan | baseline
  Thickness of different part of the cartilage of patellar measured based on axial PD images
The T2 mapping value of the patellar cartilage on 7T MRI scan | baseline
  T2 relaxation times of the patellar cartilage measured based on T2 mapping
The abnormal signal in the infrapatellar fat pad | baseline
  The exist of abnormal signal in the infrapatellar fat pad detected based on sagittal PD images

SECONDARY OUTCOMES:
Signal change of the patellar chondral before and after rehabilitation | 1 month after rehabilitation
  The correlation between abnormal change of the patellar chondral and reaction 1 month after rehabilitation
Signal change of the infrapatellar fat pad before and after rehabilitation | 1 month after rehabilitation
  The correlation between abnormal signal in the infrapatellar fat pad and reaction 1 month after rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China